CLINICAL TRIAL: NCT02276105
Title: Investigation of Psychometric Properties of the EuroQoL EQ-5D-5L in Patients With Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: Eq5d_val_cts
Record Dates: First submitted 2014-10-16; First posted 2014-10-27 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Quality of Life; EQ-5D; SF-12; Michigan Hand Questionnaire
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaires — On three time-points (Baseline, Retest, Follow-Up), each participant has to fill out the questionnaires: Michigan Hand Questionnaire, EuroQol EQ-5D-5L and the Short Form SF-12 Health Survey

SUMMARY:
The purpose of this study is to determine how appropriate and practically is the EQ-5D questionnaire in use on patients with carpal tunnel syndrome undergoing surgery along the change of quality of life.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is one of the most indications in hand surgery. To rate surgery's outcome, hand-specific instruments like the Michigan Hand Questionnaire (MHQ) are used as well as questionnaires which refers to the quality of life (QOL). In clinical daily grind, the SF-12 or the EQ-5D are common instruments to gain information about the patient's QOL. At the time, there is no current evidence available while using standardized questionnaires like the EQ-5D to capture the change in QOL in patients with CTS undergoing surgery. It would be interesting to assert that the investigation offers results about the patient's QOL and its change. Therefore, the aim of the study is to investigate the psychometric properties of the EQ-5D on patients with CTS undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* diagnosed CTS
* planned surgical decompression of the carpal tunnel
* signed informed consent

Exclusion Criteria:

* additional simultaneously performed hand surgery of the affected limb
* recurrent surgery on the already involved hand
* the other hand is already included in the study
* disease, which do not allow appropriated analysis of data like central-neurological, psychiatric or metabolic disease
* legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Schulthess Klinik (Zurich, Switzerland) with will be asked to participate on the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Quality of life measured with the EQ5D | from two weeks before surgery (Baseline) to six weeks postoperative (Follow-Up)

SECONDARY OUTCOMES:
Quality of life measured with the SF 12 | from two weeks before surgery (Baseline) to six weeks postoperative (Follow-Up)
Hand function measured with the MHQ | from two weeks before surgery (Baseline) to six weeks postoperative (Follow-Up)

CONTACTS AND LOCATIONS:
Overall Officials: Herren Daniel, Dr. med., Principal Investigator — Schulthess Klinik, Zurich, Switzerland
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Background] Marks M, Audige L, Herren DB, Schindele S, Nelissen RG, Vliet Vlieland TP. Measurement properties of the German Michigan Hand Outcomes Questionnaire in patients with trapeziometacarpal osteoarthritis. Arthritis Care Res (Hoboken). 2014 Feb;66(2):245-52. doi: 10.1002/acr.22124. PMID 23982906
- [Background] Assmus H, Antoniadis G, Bischoff C, Haussmann P, Martini AK, Mascharka Z, Scheglmann K, Schwerdtfeger K, Selbmann HK, Towfigh H, Vogt T, Wessels KD, Wustner-Hofmann M. [Diagnosis and therapy of carpal tunnel syndrome--guideline of the German Societies of Handsurgery, Neurosurgery, Neurology, Orthopaedics, Clinical Neurophysiology and Functional Imaging, Plastic, Reconstructive and Aesthetic Surgery, and Surgery for Traumatology]. Handchir Mikrochir Plast Chir. 2007 Aug;39(4):276-88. doi: 10.1055/s-2007-965464. German. PMID 17724650
- [Background] Changulani M, Okonkwo U, Keswani T, Kalairajah Y. Outcome evaluation measures for wrist and hand: which one to choose? Int Orthop. 2008 Feb;32(1):1-6. doi: 10.1007/s00264-007-0368-z. Epub 2007 May 30. PMID 17534619